CLINICAL TRIAL: NCT04735068
Title: The LIMIT KRAS Mutant NSCLC Trial: Lysosome Inhibition to Enhance MAPK Inhibition Targeting KRAS Mutant NSCLC: A Phase 2 Open Label Trial of Binimetinib and Hydroxychloroquine in Patients With Advanced KRAS Mutant Non-Small Cell Lung Cancer
Brief Title: Binimetinib and Hydroxychloroquine in Patients With Advanced KRAS Mutant Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 21520; 844511 (Other: University of Pennsylvania Office of Regulatory Affairs)
Record Dates: First submitted 2021-01-11; First posted 2021-02-02 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Cancer; KRAS Mutation-Related Tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — binimetinib; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Binimetinib and Hydroxychloroquine (Experimental): Hydroxychloroquine (HCQ)in combination with Binimetinib (B). The starting dose for HCQ will be 400mg. Tablets of HCQ are available in 200 mg strength. HCQ will be administered in divided doses (every 12 hours) with or without food.
  The starting dose of B is 45mg. B will be administered in divided doses (every 12 hours) with or without food
  Interventions: Drug: Binimetinib Pill; Drug: Hydroxychloroquine Pill

INTERVENTIONS:
Drug: Binimetinib Pill — Patients will be treated with B 45 mg two times daily and HCQ 400 mg twice daily beginning on day 1. The dose of HCQ is based on an ongoing Phase 1 trial, and may be modified in a future amendment prior to the first patient enrolled. Efforts will be made to ensure dose homogeneity throughout the trial. Treatment will be administered on an outpatient basis on a 28 day cycle
Drug: Hydroxychloroquine Pill — Patients will be treated with B 45 mg two times daily and HCQ 400 mg twice daily beginning on day 1. The dose of HCQ is based on an ongoing Phase 1 trial, and may be modified in a future amendment prior to the first patient enrolled. Efforts will be made to ensure dose homogeneity throughout the trial. Treatment will be administered on an outpatient basis on a 28 day cycle

SUMMARY:
This study will evaluate using hydroxychloroquine (HCQ) along with binimetinib as an effective method for treating cancer. All patients will receive binimetinib at a standard dose approved for other cancers. The dose of HCQ will also be fixed based on ongoing phase I studies. Eligible subjects will have lung cancer that has a mutation in a key cancer gene called KRAS, and the cancer has spread to other parts of their body.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic or incurable NSCLC
2. Presence of a non-synonymous mutation in KRAS
3. Patient must have received at least one prior systemic therapy for metastatic NSCLC or be intolerant/ineligible/refuse available therapies with known benefit
4. Ability and willingness to sign a written informed consent document
5. Age ≥18 years old
6. At least one measureable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
7. ECOG performance status 0-1
8. Adequate organ function
9. Women of childbearing potential must have a negative serum pregnancy test performed within 72hours of the first dose of study therapy. Subjects of reproductive potential must agree to use acceptable birth control methods (see Appendix B for childbearing potential).
10. Qtc < 500 mSec on EKG
11. Must be able to swallow tablets
12. Must be willing to comply with protocol procedures (including completion of diaries and outcome measures

Exclusion Criteria:

1. Currently participating in or has participated in a study of an investigational agent or anticipated use of an investigational device within 4 weeks of the first dose of study treatment.
2. Untreated symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis.
3. Prior monoclonal antibody within 4 weeks prior to enrollment, or individuals who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, non-invasive bladder tumors, or in situ cervical cancer
5. Active infection requiring systemic therapy with IV antibiotics
6. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
7. Known psychiatric or substance abuse disorders as documented in the chart that, in the opinion of the investigator, would interfere with cooperation with the requirements of the trial.
8. Pregnant or breastfeeding women
9. Anticipated receipt of any live vaccine within 30 days prior to the first dose of trial treatment.
10. Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug, or excipients or to dimethyl sulfoxide (DMSO).
11. Patients receiving cytochrome P450 enzyme-inducing anticonvulsant drugs (EIADs) (i.e.

    phenytoin, carbamazepine, Phenobarbital, primidone or oxcarbazepine) within 4 weeks of the start of the study treatment
12. Known Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (subjects with laboratory evidence of cleared HBV and/or HCV will be permitted)
13. Patients with a previously documented retinal vein occlusion.
14. History or evidence of increased cardiovascular risk including any of the following:

    * Current clinically significant uncontrolled arrhythmias. Exception: Subjects with controlled atrial fibrillation for > 30 days prior to randomization are eligible.
    * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization.
    * Ejection fraction of ≤50% as measured by echocardiography or MUGA
15. Any other conditions judged by the investigator that would limit the evaluation of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-08-21 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charu Aggarwal, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Aggarwal C, Maity AP, Bauml JM, Long Q, Aleman T, Ciunci C, D'Avella C, Volpe M, Anderson E, Jones LM, Sun L, Singh AP, Marmarelis ME, Cohen RB, Langer CJ, Amaravadi R. A Phase II Open-Label Trial of Binimetinib and Hydroxychloroquine in Patients With Advanced KRAS-Mutant Non-Small Cell Lung Cancer. Oncologist. 2023 Jul 5;28(7):644-e564. doi: 10.1093/oncolo/oyad106. PMID 37186063

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Hydroxychloroquine + Binimetinib: Hydroxychloroquine (HCQ) 400 mg twice daily Binimetinib - 45 mg twice daily
Period: Overall Study
Arm/Group | Single Arm: Hydroxychloroquine + Binimetinib
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Binimetinib and Hydroxychloroquine: Hydroxychloroquine (HCQ)in combination with Binimetinib (B). The starting dose for HCQ will be 400mg. Tablets of HCQ are available in 200 mg strength. HCQ will be administered in divided doses (every 12 hours) with or without food.
  The starting dose of B is 45mg. B will be administered in divided doses (every 12 hours) with or without food
  Binimetinib Pill: Patients will be treated with B 45 mg two times daily and HCQ 400 mg twice daily beginning on day 1. The dose of HCQ is based on an ongoing Phase 1 trial, and may be modified in a future amendment prior to the first patient enrolled. Efforts will be made to ensure dose homogeneity throughout the trial. Treatment will be administered on an outpatient basis on a 28 day cycle
  Hydroxychloroquine Pill: Patients will be treated with B 45 mg two times daily and HCQ 400 mg twice daily beginning on day 1. The dose of HCQ is based on an ongoing Phase 1 trial, and may be modified in a future amendment prior to the first patient enrolled. Efforts will be made to ensure dose homogeneity throughout the trial. Treatment will be administered on an outpatient basis on a 28 day cycle
Arm/Group | Binimetinib and Hydroxychloroquine
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 64 [52 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Hydroxychloroquine + Binimetinib
Number analyzed (Participants) | 9
Participants | 9

2. Primary Outcome: Number of Patients With Adverse Events
Description: as assessed by CTCAE v5.0
Time Frame: 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib and Hydroxychloroquine
Number analyzed (Participants) | 9
Participants | 9

3. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib and Hydroxychloroquine
Number analyzed (Participants) | 9
Participants | 1

4. Secondary Outcome: Overall Survival (OS)
Time Frame: 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Hydroxychloroquine + Binimetinib
Number analyzed (Participants) | 9
Participants | 1

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Single Arm: Hydroxychloroquine + Binimetinib
All-Cause Mortality (participants affected / at risk) | 1/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm: Hydroxychloroquine + Binimetinib (N=9)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm: Hydroxychloroquine + Binimetinib (N=9)
Rash (Skin and subcutaneous tissue disorders) | 6 (14)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
ALT Increase (Investigations) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
AST Increased (Investigations) | 1 (4)
Collitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Dry Skim (Skin and subcutaneous tissue disorders) | 1 (1)
Edema Face (General disorders) | 2 (2)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Subfoveal Serous Detachment (Eye disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Under Tongue Swelling (General disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Retinal Detachment (Eye disorders) | 1 (1)
Vomitting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT04735068/Prot_SAP_000.pdf